CLINICAL TRIAL: NCT00001536
Title: Issues Surrounding Prenatal Genetic Testing for Achondroplasia
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960123; 96-HG-0123
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-08

CONDITIONS: Achondroplasia; Dwarfism
Keywords: Disability; Dwarfism; Ethics in Genetic Counseling; Quality of Life; Reproductive Issues; Support Groups; Achondroplasia
MeSH Terms: conditions — Achondroplasia; Dwarfism

SUMMARY:
Since the gene responsible for achondroplasia was identified in 1994, it has become possible to test for achondroplasia prenatally. Moreover, prenatal genetic testing for achondroplasia is relatively simple and is highly likely to be informative for any couple seeking testing. Four diagnostic laboratories in the U.S. are currently performing prenatal genetic testing for achondroplasia. Before prenatal genetic testing for achondroplasia becomes more widely available, however, it is essential that we learn more about the lives of affected individuals and their families, the implications of offering testing for achondroplasia, and the education and the counseling needs of this community. Personal interviews and stories have been published and discussed at national meetings (Ablon 1984). We conducted a pilot telephone interview survey of 15 individuals with achondroplasia. What is needed now is a large scale quantitative study of the community of little people and their families. To meet this need, we have developed a survey tool to analyze family relationships, quality of life, tendencies toward optimism or pessimism, information-avoiding or information-seeking behaviors, social support, involvement in Little People of America Inc. (LPA), self-esteem, sociodemographics and views on achondroplasia, religiousness, reproductive and family plans, genetic testing, and abortion. The self-administered survey will be completed nationally by a sample of persons with achondroplasia and their family members.

DETAILED DESCRIPTION:
Since the gene responsible for achondroplasia was identified in 1994, it has become possible to test for achondroplasia prenatally. Moreover, prenatal genetic testing for achondroplasia is relatively simple and is highly likely to be informative for any couple seeking testing. Four diagnostic laboratories in the U.S. are currently performing prenatal genetic testing for achondroplasia. Before prenatal genetic testing for achondroplasia becomes more widely available, however, it is essential that we learn more about the lives of affected individuals and their families, the implications of offering testing for achondroplasia, and the education and the counseling needs of this community. Personal interviews and stories have been published and discussed at national meetings (Ablon 1984). We conducted a pilot telephone interview survey of 15 individuals with achondroplasia. What is needed now is a large scale quantitative study of the community of little people and their families. To meet this need, we have developed a survey tool to analyze family relationships, quality of life, tendencies toward optimism or pessimism, information-avoiding or information-seeking behaviors, social support, involvement in Little People of America Inc. (LPA), self-esteem, sociodemographics and views on achondroplasia, religiousness, reproductive and family plans, genetic testing, and abortion. The self-administered survey will be completed nationally by a sample of persons with achondroplasia and their family members.

ELIGIBILITY:
Adult individuals of either gender with achondroplasia and their first degree relatives (both short and average statured) of all ethnic and cultural backgrounds.

No short-statured persons with conditions other than achondroplasia.

No average-statured family members of short statured persons with conditions other than achondroplasia.

No minors less than 18 years of age.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000
Dates: Start 1996-08; Study Completion 2000-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute (NHGRI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bellus GA, Escallon CS, Ortiz de Luna R, Shumway JB, Blakemore KJ, McIntosh I, Francomano CA. First-trimester prenatal diagnosis in couple at risk for homozygous achondroplasia. Lancet. 1994 Nov 26;344(8935):1511-2. doi: 10.1016/s0140-6736(94)90332-8. No abstract available. PMID 7968151
- [Background] Bellus GA, Hefferon TW, Ortiz de Luna RI, Hecht JT, Horton WA, Machado M, Kaitila I, McIntosh I, Francomano CA. Achondroplasia is defined by recurrent G380R mutations of FGFR3. Am J Hum Genet. 1995 Feb;56(2):368-73. PMID 7847369
- [Background] Elejalde BR, de Elejalde MM, Hamilton PR, Lombardi JM. Prenatal diagnosis in two pregnancies of an achondroplastic woman. Am J Med Genet. 1983 Jul;15(3):437-9. doi: 10.1002/ajmg.1320150308. PMID 6881210